CLINICAL TRIAL: NCT01733394
Title: Equivalence Among Antiepileptic Drug Generic and Brand Products in People With Epilepsy: Single-Dose 6-Period Replicate Design (EQUIGEN Single-Dose Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: American Epilepsy Society (Other); Epilepsy Foundation (Other)
Responsible Party: Principal Investigator, Michael Privitera, Director Cincinnati Epilepsy Center, University of Cincinnati
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: EQUIGEN Single Dose Protocol; 005-1005 (Other Grant/Funding Number: 005-1005)
Record Dates: First submitted 2012-11-02; First posted 2012-11-27 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Epilepsy
Keywords: Epilepsy; Generic
MeSH Terms: conditions — Epilepsy | interventions — Lamotrigine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Generic A - Generic B - Brand - Generic A - Brand - Generic B (Experimental): Sequence 1
  Interventions: Drug: Lamotrigine Generic "A" Lamotrigine Generic "B" Lamotrigine "Brand"; Drug: lamotrigine
- Generic B - Brand - Generic A - Generic B - Generic A - Brand (Experimental): Sequence 2
  Interventions: Drug: Lamotrigine Generic "A" Lamotrigine Generic "B" Lamotrigine "Brand"; Drug: lamotrigine
- Brand - Generic A - Generic B - Brand - Generic B- Generic A (Experimental): Sequence 3
  Interventions: Drug: Lamotrigine Generic "A" Lamotrigine Generic "B" Lamotrigine "Brand"; Drug: lamotrigine

INTERVENTIONS:
Drug: Lamotrigine Generic "A" Lamotrigine Generic "B" Lamotrigine "Brand"
  Other Names: Lamotrigine
Drug: lamotrigine

SUMMARY:
The United States Food and Drug Administration (FDA) has specific rules which generic drug companies must follow to get a generic copy of a seizure medication approved. Currently, FDA approves generic drugs by requiring studies on normal volunteers who don't have epilepsy and who take just one dose of the generic drug followed by a series of blood tests. Some people with epilepsy and their physicians have complained about side effects or loss of seizure control when taking generic drugs, but no one knows if these complaints are truly because of problems with the generic drugs.

This research is to determine whether several different generic versions and the brand version of the medication lamotrigine perform in a similar way when given to people with epilepsy.

The study drug Lamictal® (lamotrigine) and both of the generic forms of lamotrigine to be tested are approved by the FDA for the treatment of seizures.

DETAILED DESCRIPTION:
The study proposed in this protocol will determine if bioequivalence testing performed for the FDA translates into similar bioequivalence in a population of people with epilepsy when switching among different generics of the anti-epileptic drug (AED). Based on a variety of pharmacokinetic (PK) data and clinical reports of concern, the example anti epilepsy drug (AED) used for this study will be lamotrigine (LTG).

In this single dose study, people with epilepsy taking AEDs, but not currently taking the test medication, lamotrigine, will be studied. We will use an order-randomized three-sequence six-period replicate design with the two most disparate generics studied in two replicate periods each and the brand (reference) product studied in two additional periods. A standard single dose of the test drug (lamotrigine 25mg) will be administered under controlled conditions (fasting with subsequent standardized meals) with a 12-hour in-facility blood sample collection followed by a collection every 24 hours for a total of a 96 hour sample collection that will be used to establish the pharmacokinetic measures of Cmax, AUC96 and AUC∞. Each period will be separated by at least a 12 day washout interval.

The replicate studies will be used to determine the intra-individual variability of the pharmacokinetic responses of the brand and the two generic products, as well as subject-by-formulation interaction variances. The data will also be used to calculate simultaneously all parameters that are needed to compare the 3 products in average and individual bioequivalence and outlier analyses. The differences between the disparate generics will be used to establish if the current standards translate to equivalence within the limits of the brand intra-subject variation.

The factors we will use to determine the most disparate generics include the results from the in vivo data from the ABE studies submitted to the FDA in the ANDA and in vitro chemical assay (potency) and dissolution data performed on several currently available lots. The intent is to study the specific lot of the generic product predicted to result in the lowest levels and compare it to the specific lot from another generic product predicted to result in the highest levels. Similarly, if multiple lots of the brand products are available, we will perform in vitro testing to establish the most desirable lot to study.

Factors that alter metabolism, including concomitant AEDs that may have hepatic enzyme induction effects will be tracked but not excluded, as long as the dose remains constant, as the goal is to reproduce the 'real life' situation as closely as possible within the practical limits of funding and study size. Subjects receiving valproate as concomitant medication will be excluded because the prolongation of half life would not allow LTG to reliably be completely cleared by 13 days. The criteria that establish an enriched population will also be tracked and used in a secondary analysis, but will not be used as an inclusion requirement. The enriched population is defined as people who experienced an otherwise unexplained increase in seizures or adverse effects, or a substantial change in AED level after a switch in AED products.

The discovery of any subject-by-formulation interaction outliers (i.e. subjects with differential pharmacokinetic reactions to a pair of formulations) will raise considerable concerns about equivalence. Recently established methods in the statistical analysis of outliers in crossover studies will be used to determine if any outliers are present.

Qualified subjects will be screened and upon fulfilling inclusion/exclusion criteria and signing the informed consent will be enrolled in the study and enter the randomization phase (2-30 days). Subjects will be randomized according to a sealed allocation list that will be balanced for sequence and provided to each site prior to the first subject enrollment. Subjects that withdraw prior to completing the third period will be replaced in a randomized manner. The randomization list will be generated by the study statistical group. There are six test periods in three sequences for a sequence-randomized study. During two test periods subjects will receive a single dose of the brand AED and during the other four test periods subjects will receive a single dose from one of the two investigated generics (each twice). The single doses will be administered in the fasting state during an in-facility 12-hour pharmacokinetic session to collect samples to determine Cmax and AUCs. Four additional samples will be drawn at 24, 48, 72, and 96 hours after the dose as an outpatient (making each pharmacokinetic test last for 4 days). Each in-facility pharmacokinetic testing will be separated by a 12-23 day washout period; consistent washout periods of 14 days will be preferred. A final follow-up phone evaluation will be conducted 12-16 days (target 14 days) after the last dose. During the study the subjects will continue their usual concomitant medications, including AEDs, without change.

Investigators will compare the AED levels as measured by Cmax and AUC in each group using average bioequivalence (ABE) and individual bioequivalence (IBE) criteria. Average bioequivalence will be established if the 90% confidence intervals of the geometric mean of Cmax and AUCs for the most disparate generic products compared to each other are entirely within the 80%-125% range (the FDA criteria for bioequivalence) using the two one-sided standard analyses. Otherwise the products will be considered to not be bioequivalent. Similarly, the products will be considered to not be bioequivalent if the criteria for IBE for each generic product compared to the brand product are not met.

Study Population: Approximately 54 subjects (45 subjects to completion).

Number of centers: 3 sites enrolling approximately 18 subjects each.

Duration of study: Approximately 1 year.

ELIGIBILITY:
Inclusion Criteria

Eligible subjects must satisfy the criteria below at the time of enrollment:

1. 18 years or older.
2. BMI not less than 18.5 and weight not less than 110 pounds.
3. Not donated blood within the past 56 days before the first pharmacokinetic testing.
4. Agrees not to donate blood at any time during the trial and for 56 days after the final PK in-facility admission.
5. Has epilepsy for at least one year based on site PIs assessment.
6. Taking at least one AED, which is not the study medication (lamotrigine).
7. No changes in AED regimen for at least 28 days prior to first pharmacokinetic testing.
8. Have the ability to understand the informed consent form and be willing to provide informed consent.
9. Willing to remain on same AED regimen through entire study. Subjects will be responsible to supply all of their concomitant medications (except for the study medication, lamotrigine).
10. Willing to stay approximately 14 hours in the research facility on six separate occasions for pharmacokinetic testing.
11. Willing to fast overnight and the morning of each of the six pharmacokinetic testing sessions.
12. Willing to have at least 23 blood samples collected during the pharmacokinetic testing including the in-facility session and each of the following four mornings for 96 hours post the study medication dose to complete the sample collection for each of the 6 periods. The in-facility blood collections will mainly be performed using an inserted catheter. In the event of difficulty with the catheter, samples may be drawn by venipuncture. The outpatient collections will be drawn by venipuncture. The total amount of blood during each PK session will be equal to about 14 teaspoons (66.5 milliliters). The total amount of blood drawn throughout the entire study will be about 96 teaspoons (478.5 milliliters) or less. For reference, this amount is approximately equal to the quantity of blood drawn during a standard blood donation by the Red Cross.
13. Willing to completely abstain from alcohol consumption for at least 24 hours prior to each pharmacokinetic testing admission until after the last sample is drawn for each period (~96 hours after the initial dose at each pharmacokinetic admission). We encourage no or minimal alcohol use throughout the study, but alcohol is not restricted at other times.
14. Willing to remain on a consistent regimen of concomitant medications including over-the-counter drugs and herbal drugs, if they are being used and deemed to possibly affect the metabolism of the study medication.
15. Willing to not eat grapefruit or drink grapefruit juice through the duration of the study.
16. If a tobacco user, willing to continue with the same pattern of tobacco use, except that no tobacco use is permitted during the PK facility admissions of approximately 14 hours (includes all tobacco products).
17. Willing to complete the subject diary as outlined in the protocol.
18. Willing to adhere to all other protocol requirements as outlined in the informed consent document.
19. Females must be either of non-childbearing potential (defined as having undergone surgical sterilization or postmenopausal (greater than 50 years old and amenorrhea for greater than or equal to 12 months) or must be using at least one acceptable method of contraception as follows:

    1. Double-barrier method (e.g. condom plus spermicide, condom plus diaphragm with spermicide)
    2. Hormonal contraceptive treatment (progesterone only agents - use of any agents containing estrogen are an exclusion for the lamotrigine testing)
    3. Intrauterine Device (IUD)
    4. Monogamous relationship with a vasectomized partner
    5. Abstinent for 8 weeks prior to and throughout the study.
20. Subject must be at least 28 days from last participation in any other study.

Exclusion Criteria

1. Progressive CNS disorder that could influence adverse effects or seizure control.
2. Known medication non-adherence. Non-adherence is assessed by the investigator based on the procedures defined in the manual of procedures.
3. Taking the study medication (lamotrigine) within 28 days of enrollment.
4. Use of valproate (as divalproex sodium or valproic acid), any form of estrogens, rifampin, orlistat, felbamate or sertraline within 28 days of study entry.
5. Subject has a history of alcohol or substance abuse within 1 year prior to screening for study participation, or is currently using alcohol, drugs of abuse, or any prescribed or over-the-counter medication in a manner, which, in the opinion of the Investigator, indicates abuse.
6. History of psychogenic seizures within the past 2 years.
7. Any clinically significant psychiatric illness or psychological or behavioral problem which, in the opinion of the investigator, could interfere with the subject being able to participate in the study or comply with the study requirements. .
8. Any clinically significant laboratory abnormality or illness which, in the opinion of the investigator, could interfere with the conducting or interpretation of the study or put the subject at risk.
9. History of allergic reaction with past use of the study medication (lamotrigine).
10. More than two allergic reactions (actual allergy, not medication intolerance) to an AED or one serious hypersensitivity reaction to an AED.
11. History of adverse effect associated with past use of the study medication (lamotrigine) which, in the opinion of the investigator, could pose substantial risk to the subject if it occurred during the trial.
12. Pregnant or lactating within 56 days of enrollment.
13. Unstable seizure control that makes AED changes likely during the course of the study.
14. Use of rescue AEDs (e.g. benzodiazepines) during more than two weeks of the 2 months prior to enrollment.
15. Subject is in the process of quitting smoking within 28 days of study entry or plans to quit smoking during the period of time the study will be conducted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2012-12-12 (Actual); Primary Completion 2016-09-26 (Actual); Study Completion 2016-09-26 (Actual)

PRIMARY OUTCOMES:
Bioequivalence for generic 1 compared to generic 2 | 18 months
  To determine if Cmax or AUC are significantly different in the high generic product compared to the low generic product taking one as the reference and the other as the test product. Bioequivalence will be established per the current FDA ABE criteria if the 90% confidence interval of the geometric mean of Cmax and AUC for the high generic product compared to the low generic product are entirely within the 80%-125% range using the two one-sided standard analyses

SECONDARY OUTCOMES:
Intra-subject variances | 18 months
  To measure the intra-subject variances of the investigated REFERENCE (BRAND) AND generic products, as well as subject-by-interaction variances, by using two replicate periods for THE REFERENCE PRODUCT AND TWO REPLICATE PERIODS FOR each generic product. These estimated variances will be used to investigate individual bioequivalence and detect subject-by-formulation interaction outliers

OTHER OUTCOMES:
Individual Bioequivalence | 18 months
  To examine individual bioequivalence by comparing the BRAND TO EACH OF THE two generic products. Individual bioequivalence (IBE) will be determined using the FDA 2001 guidance criteria. To determine the number of subjects who are outliers and to identify these subjects for potential further study.
Bioequivalence for subjects receiving inducers compared to not receiving inducers | 18 months
  To compare the REFERENCE/generic and generic1 /generic2 ratios for Cmax and AUC in subjects on a concomitant enzyme inducing AED compared to subjects not on a concomitant enzyme AED
Bioequivalence by gender | 18 months
  To compare the REFERENCE/generic and generic1/generic2 ratios for Cmax and AUC in male subjects compared to female subjects
Bioequivalence in enriched population | 18 months
  To compare the REFERENCE/generic and generic1/generic2 ratios for Cmax and AUC in the population of subjects who had reported loss of seizure control or unanticipated adverse effects after a generic switch.

CONTACTS AND LOCATIONS:
Overall Officials: Michael D. Privitera, MD, Principal Investigator — University of Cincinnati; Michel J Berg, MD, Principal Investigator — University of Rochester
Locations (8):
- United States (8):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Drake University, Des Moines, Iowa
  - University of Iowa, Iowa City, Iowa
  - University of Kansas, Kansas City, Kansas
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Rochester Medical Center, Rochester, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - University of Wisconsin-Madison, Madison, Wisconsin

REFERENCES:
- [Derived] Berg M, Welty TE, Gidal BE, Diaz FJ, Krebill R, Szaflarski JP, Dworetzky BA, Pollard JR, Elder EJ Jr, Jiang W, Jiang X, Switzer RD, Privitera MD. Bioequivalence Between Generic and Branded Lamotrigine in People With Epilepsy: The EQUIGEN Randomized Clinical Trial. JAMA Neurol. 2017 Aug 1;74(8):919-926. doi: 10.1001/jamaneurol.2017.0497. PMID 28654954